CLINICAL TRIAL: NCT00335309
Title: Effectiveness of Maxillary Sinus Saline Irrigation in Conjunction With Systemic Antibiotic Therapy Versus Systemic Antibiotic Therapy Alone in the Management of Chronic Rhinosinusitis, a Prospective Randomized Controlled Trial
Brief Title: Maxillary Sinus Irrigation in the Management of Chronic Rhinosinusitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohad Ronen (Other)
Responsible Party: Sponsor-Investigator, Ohad Ronen, ENT Physician, Carmel Medical Center
Organization: Carmel Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ENT-1/2005; 20051031 (Other: CMC 09-0072)
Record Dates: First submitted 2006-06-08; First posted 2006-06-09 (Estimated); Last update posted 2013-10-08 (Estimated); Status verified 2013-10

CONDITIONS: Sinusitis
Keywords: chronic rhinosinusitis; sinus irrigation
MeSH Terms: conditions — Sinusitis | interventions — Amoxicillin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): The Investigational arm is treated with sinus irrigation with normal saline 0.9% and intravenous antibiotics of Augmentin 1 gram 3 times a day for 4 days, and then per os (PO) Augmentin 875mg twice a day (BID) for another 10 days. The treatment is done while the patient is admitted to the otolaryngology - head and neck surgery department.
  Interventions: Procedure: Maxillary Sinus Irrigation
- 2 (Active Comparator): The control arm is treated with the same intravenous antibiotics of Augmentin 1 gram 3 times a day for 4 days, and then per os (PO) Augmentin 875mg twice a day (BID) for another 10 days. There is no sinus irrigation with normal saline for this arm. The treatment is done while the patient is admitted to the otolaryngology - head and neck surgery department.
  Interventions: Drug: IV Amoxicillin and Clavulanate acid

INTERVENTIONS:
Procedure: Maxillary Sinus Irrigation — Twice a day irrigation with 100cc saline for 4 days
  Arms: 1
Drug: IV Amoxicillin and Clavulanate acid — IV Amoxycillin and Clavulanate 1 Gram TID for 4 days.
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the effectiveness of maxillary sinus saline irrigation in conjunction with systemic antibiotic therapy versus systemic antibiotic therapy alone in the management of chronic rhinosinusitis, a prospective randomized controlled trial.

DETAILED DESCRIPTION:
Effectiveness of maxillary sinus saline irrigation in conjunction with systemic antibiotic therapy versus systemic antibiotic therapy alone in the management of chronic rhinosinusitis. A prospective randomized controlled trial is being conducted in Carmel Medical Center, Haifa, Israel. Patients are being randomized into one of two arms. One arm receives sinus irrigation with saline in conjunction with IV antibiotics, the control arm receives the same regimen of IV antibiotics without the sinus irrigation. Quality of life, CT scans and nasal endoscopy parameters are collected before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Chronic (over 3 months) maxillary and ethmoidal rhinosinusitis (verified by a CT scan)
* Over 18 years of age
* Signed informed consent
* Not participating in another clinical study

Exclusion criteria:

* A previous sinonasal surgery or craniofacial trauma
* Isolated frontal or sphenoidal sinusitis
* Immunosuppressed (diabetes, cancer, etc.)
* Craniofacial deformity
* Allergic fungal sinusitis
* Nasal polyposis
* Rhinosinusitis of dental origin
* Bleeding tendency (e.g., chronic coumadin treatment)
* Patients participating in other clinical study
* Patients with penicillin allergy
* Patients with Augmentin resistant bacteria in cultures

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2005-10; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
CT Scoring | on recruiting and follow-up

SECONDARY OUTCOMES:
Quality of life Questionaire | on recruiting and follow-up
Nasal Endoscopy score | upon recruiting and follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Ohad Ronen, MD, Principal Investigator — ENT Department, Carmel Medical Center, Haifa
Locations (1):
- Carmel MC, Haifa, Israel

REFERENCES:
- [Background] Benninger MS, Sedory Holzer SE, Lau J. Diagnosis and treatment of uncomplicated acute bacterial rhinosinusitis: summary of the Agency for Health Care Policy and Research evidence-based report. Otolaryngol Head Neck Surg. 2000 Jan;122(1):1-7. doi: 10.1016/S0194-5998(00)70135-5. PMID 10629474
- [Background] Gliklich RE, Metson R. The health impact of chronic sinusitis in patients seeking otolaryngologic care. Otolaryngol Head Neck Surg. 1995 Jul;113(1):104-9. doi: 10.1016/S0194-59989570152-4. PMID 7603703
- [Background] Benninger MS, Appelbaum PC, Denneny JC, Osguthorpe DJ, Stankiewicz JA. Maxillary sinus puncture and culture in the diagnosis of acute rhinosinusitis: the case for pursuing alternative culture methods. Otolaryngol Head Neck Surg. 2002 Jul;127(1):7-12. doi: 10.1067/mhn.2002.124847. PMID 12161724